CLINICAL TRIAL: NCT00524797
Title: Profonycia - Honey for Improving Quality of Patient's Life Receiving Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HP 7-260 S
Record Dates: First submitted 2007-09-02; First posted 2007-09-05 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-09

CONDITIONS: Myelosuppression
Keywords: Myelosuppression,; chemotherapeutic agents,; leucopenia,; thrombocytopenia,; Profonycia
MeSH Terms: conditions — Leukopenia; Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Main (Active Comparator): 50 patients will receive Profonycia 5 gr/day PO for 7 days
  Interventions: Dietary Supplement: Profonycia

INTERVENTIONS:
Dietary Supplement: Profonycia

SUMMARY:
Myelosuppression (bone marrow suppression) is the most important toxic side effect of the majority of chemotherapeutic agents and typically is the dose limiting factor. Death occurring after chemotherapy usually results either from infection related to drug induced leucopenia or from bleeding related to thrombocytopenia. Colony stimulating factors (CSFs) are widely used in the treatment of chemotherapy induced neutropenia. The same Erythropoetines are used in the treatment of chemotherapy induced anemia. Both treatments are expensive and have several side effects.

In our previous stud (1) we found a special kind of honey: Life-Mel Honey to reduce the incidence of chemotherapy induced pancytopenia and improving quality of life.

The aim of the recent planed study is to provide prophylactic and protective treatment against neutropenia reducing the need for secondary CSF administration in patients receiving chemotherapy along with a natural and non expensive honey: Profonycia.

This honey which is expressed in Kibutz Shamir in Upper Galliee seems promising and easy for administration: given 5 gr/day per os for 7 days from the administration of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years old or elder receiving chemotherapy 1/2-3 weeks

Exclusion Criteria:

Patients below 18 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Zidan Jamal, Prof, Principal Investigator — Ziv MC
Locations (2):
- Israel (2):
  - Oncology Unit, Ziv MC, Safed
  - Oncology Unit, Safed

REFERENCES:
- [Background] Zidan J, Shetver L, Gershuny A, Abzah A, Tamam S, Stein M, Friedman E. Prevention of chemotherapy-induced neutropenia by special honey intake. Med Oncol. 2006;23(4):549-52. doi: 10.1385/MO:23:4:549. PMID 17303914